CLINICAL TRIAL: NCT05218031
Title: Acceptance and Commitment Group Therapy for Unaccompanied Minors: A Pilot Study
Brief Title: Acceptance and Commitment Group Therapy for Unaccompanied Minors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Maria Karekla, Associate Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K3_K1_1
Record Dates: First submitted 2021-12-10; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Post Traumatic Stress Disorder; Depression; Anxiety Disorders
Keywords: Unaccompanied Refugee Minors; Acceptance and Commitment Therapy; Child/Adolescent Mental Health; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: A two-arm randomised trial will be conducted (brief ACT-based intervention vs. waiting-list control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Intervention (Experimental): 5-week ACT Group Intervention based on the Self-Help Booklet by the World Health Organization "Doing What Matters in Times of Stress: An Illustrated Guide".
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control group (No Intervention): Waiting-list

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — A 90-120 minute 5-week group intervention for unaccompanied minors. Each week there will be a different focus. Week 1: Grounding, Week 2: Unhooking, Week 3: Values, Week 4: Self-compassion, Week 5: Making room for unwanted thoughts and feelings.
  Arms: ACT Intervention

SUMMARY:
Unaccompanied minors (UM) are considered to be a highly vulnerable refugee subgroup. Research has indicated that UM experience traumatic events and consequently develop high levels of psychopathology. Post-traumatic stress disorder is the most prevalent diagnosis, followed by depression, anxiety disorders as well as traumatic grief and conduct problems. Acceptance and Commitment Therapy (ACT) may be particularly suited to the treatment of survivors of trauma and with vulnerable refugee groups such as UM. A 5-week ACT group intervention will be carried out and its feasibility in UM will be explored along with its effect on mental health. The ACT group intervention will be based on a Self-Help Booklet by the World Health Organization "Doing What Matters in Times of Stress: An Illustrated Guide". Following the 5-week ACT group intervention, focus groups with participants will be carried out to examine its acceptability and will be analysed qualitatively, using thematic analysis.

DETAILED DESCRIPTION:
The hypotheses of the study are as follows:

1. The ACT group intervention will lead to increases in UM psychological well-being and quality of life compared to a waiting-list (WL) control group. This includes improvements in post-traumatic stress symptoms, depression, anxiety, stress, and sleep difficulties. (Primary outcomes).
2. The UM receiving the ACT group intervention will demonstrate improvements in their prosocial behaviour compared to the WL control group. (Primary outcomes).
3. At post-intervention, UM receiving the ACT group intervention will have enhanced psychological flexibility compared to the WL control group. It is predicted that there will be decreased experiential avoidance and cognitive fusion, coupled with increases in values-driven committed action, present moment awareness and self-as-context. (Secondary outcomes).
4. At the 1-month and 3-month follow-up time points, the UM receiving the ACT group intervention will have retained the improvements from the treatment (i.e., increased psychological wellbeing, enhanced psychological flexibility, augmented prosocial behaviour) compared to the WL control group. Additionally, it is predicted that UM who completed the ACT group intervention will not only have sustained the benefits observed directly post-intervention but will in fact keep making progress at follow-up time points compared to the WL control group.

From the qualitative analysis, the investigators presume to provide critical insights as to what is perceived acceptable and culturally appropriate treatment for this population.

ELIGIBILITY:
Inclusion Criteria:

* Unaccompanied refugee minors living in sheltered accommodation in Cyprus.
* No specific diagnosis required to take part in the study.
* No specific cultural background required.
* Minors who provide consent.

Exclusion Criteria:

- Presence of active psychosis.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in 'Quality of Life': KIDSCREEN-27 (Ravens-Sieberer et al., 2007). | Pre-intervention, Post-intervention (at 5 weeks), 1-month follow-up, 3-months follow-up
  This is a 27-item instrument that consists of five dimensions of quality of life: physical well-being (5 items), psychological well-being (7 items), autonomy and relationship with parents (7 items), peers and social support (4 items), and school environment (4 items). The questions concern the last seven days and answers are given on a five-point Likert scale ('Not at all, slightly, moderately, very, extremely' or 'never, seldom, quite often, very often, always'). Higher scores on the KIDSCREEN-27 reflect higher quality of life and wellbeing. Internal consistency of this scale was considered satisfactory (Cronbach's alpha= >.70).
Change in 'The Depression, Anxiety and Stress Scale' (DASS-21; Lovibond & Lovibond, 1995; Antony, Bieling, Cox, Enns, & Swinson., 1998). | Pre-intervention, Post-intervention (at 5 weeks), 1-month follow-up, 3-months follow-up
  This scale includes 21 items and will be used to assess for symptoms of depression, anxiety and stress in our sample. The Depression scale assesses hopelessness, low self-esteem, and low positive affect. The Anxiety scale assesses autonomic arousal, physiological hyperarousal, and the subjective feeling of fear. The Stress scale items assess tension, agitation, and negative affect. There are seven items per scale and participants must rate their past week on a Likert-type scale (0-3). Higher scores indicate higher levels of depression, stress and anxiety. Cronbach's alphas indicating high internal consistency for Depression .94, Anxiety .84 and Stress .91.
Change in 'The Child Revised Impact of Events Scale' (CRIES-8; Perrin, Meiser-Stedman, & Smith., 2005). | Pre-intervention, Post-intervention (at 5 weeks), 1-month follow-up, 3-months follow-up
  This scale will be used to assess for any post-traumatic stress symptoms. The total number of items in the scale are 8 items. Four of the items assess intrusion (intrusive thoughts, feelings) and the remaining four items assess avoidance (avoidance of situations, feelings). The items are scored on a 4- point scale, where higher scores indicate higher levels of intrusion or avoidance. The CRIES-13 (Smith, Perrin, Dyregov, & Yule, 2003) was found to have high internal consistency (Cronbach's alpha= 0.80). Sensitivity (i.e., the probability that someone with a diagnosis of PTSD will screen positive) was found to be .94-1.0. Specificity (i.e., the probability that someone without a diagnosis of PTSD will screen negative) was found to be .59-.71. The overall efficiency rate of the CRIES-8 is 75-82.7%.
Change in 'Strengths and Difficulties Questionnaire' (SDQ; Goodman, 1997; 2001). | Pre-intervention, Post-intervention (at 5 weeks), 1-month follow-up, 3-months follow-up
  This questionnaire consists of 25 items divided into five subscales with 5 items each: Emotional difficulties, Conduct problems, Hyperactivity/inattention, Peer problems and Prosocial behaviour. Each item is scored on a 3-point scale (0= 'not true', 1='somewhat true', and 2= 'certainly true'). Subscale scores are calculated by summing scores on relevant items (after recoding reversed items). Higher scores on the prosocial behaviour subscale indicate strengths, whilst higher scores on the other four subscales indicate difficulties. A total difficulties score is computed by summing the scores on all five subscales (range 0-40). Reliability of this scale is satisfactory as assessed by internal consistency (Cronbach's alpha=0.73), cross-informant correlation (mean= 0.34), and retest stability after 4 to 6 months (mean= 0.62).

SECONDARY OUTCOMES:
Change in the ACT Process Measure: PsyFlex (Gloster et al., 2021). | Pre-intervention, throughout study completion 5 weeks, 1-month follow-up, 3-months follow-up
  This is an 8-item self-report questionnaire which assesses the process of psychological flexibility. Each item is rated on a five-point scale from 1 (very often) to 5 (very rarely).

OTHER OUTCOMES:
Treatment Adherence Measure: ACT Fidelity Measure (ACT-FM; O'Neill et al., 2019). | up to 5 weeks
  This questionnaire consists of 25 items which capture four key areas within ACT: Therapist Stance (7 items), Open Response Style (6 items), Aware Response Style (6 items) and Engaged Response Style (6 items). Within each area there are items to score the therapist's behaviour as ACT consistent and ACT inconsistent. Scoring is rated on a 4-point scale from 0-3 (0= 'This behaviour never occurred', 1= 'Therapist rarely enacts this behaviour', 2= 'Therapist sometimes enacts this behaviour', 3= 'Therapist consistently enacts this behaviour'). Within 'Engaged response style' for instance, "Therapist gives the client opportunities to clarify their own values" would be considered ACT consistent, "Therapist imposes their own, other's or society's values upon the client" would be considered ACT inconsistent. A total score can be calculated for each subscale as well as a total ACT consistent score and total ACT inconsistent score. Inter-rater reliability was deemed moderate to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Karekla, Ph.D., Principal Investigator — University of Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University Clinical Laboratory Website — http://www.ucy.ac.cy/acthealthy/en/